CLINICAL TRIAL: NCT06523790
Title: Comparative Study on the Effects of Brisk Walking and Yoga on Glucose and Lipid Metabolism and Neurocognitive Function in Adults: A Randomized Controlled Trial
Brief Title: The Impact of Exercise Methods on Human Body Functions and Metabolism
Acronym: EXMET-BW&Y
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhoukou Normal University (Other)
Responsible Party: Principal Investigator, Jin Li, instructor, Zhoukou Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhoukouNU-001
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome
Keywords: Yoga, Walking, Exercise, Body Composition, Metabolic Health
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Participants in this group will undergo 90-minute yoga sessions, 3 times per week, for 8 months. The yoga intervention includes a combination of asanas (postures), pranayama (breathing exercises), and meditation designed to improve flexibility, strength, and mental well-being.
  Interventions: Behavioral: Yoga
- Walking Group (Experimental): Participants in this group will engage in one-hour fast-paced walking sessions, 6 times per week, for 8 months. The walking intervention is designed to improve cardiovascular fitness, endurance, and support weight loss.
  Interventions: Behavioral: Brisk walking

INTERVENTIONS:
Behavioral: Yoga — Participants in the yoga group will attend 90-minute yoga sessions, 3 times per week, for 8 months. The sessions will include a combination of asanas (postures), pranayama (breathing exercises), and meditation.
  Arms: Yoga Group
Behavioral: Brisk walking — Participants in the brisk walking group will engage in one-hour fast-paced walking sessions, 6 times per week, for 8 months. The walking regimen is designed to improve cardiovascular fitness, endurance, and support weight loss.
  Arms: Walking Group

SUMMARY:
The objective of this study is to compare the effects of 8 months of yoga and walking exercise training on weight-related body fat and metabolic biomarkers in women. Participants will be randomly assigned to either a yoga group or a walking group. The yoga group will undergo 90-minute sessions, 3 times per week, while the walking group will engage in one-hour sessions, 6 times per week. Physical and metabolic markers will be measured at baseline and after 8 months of intervention.

DETAILED DESCRIPTION:
This randomized controlled trial aims to investigate the differential impacts of yoga and walking exercise training on weight-related body fat and metabolic biomarkers in women over an 8-month period. The study will recruit women aged 18-65 years, who will be randomly assigned to either a yoga group or a walking group.

Yoga Group: Participants in the yoga group will attend 90-minute yoga sessions, 3 times per week.

Walking Group: Participants in the walking group will engage in one-hour fast-paced walking sessions, 6 times per week.

Outcome Measures: Physical and metabolic markers will be assessed at baseline and after 8 months of exercise intervention. The primary outcomes will include changes in body weight, BMI, visceral fat, and basal metabolism. Metabolic biomarkers such as serum leptin, glucose, total cholesterol (TC), apolipoprotein A (APOA), and apolipoprotein B (APOB) will also be measured.

Participants will be monitored for adherence to the exercise protocol and any adverse events throughout the study. Data will be collected during the intervention, and analyzed to determine the differential effects of yoga and walking on the measured outcomes.

The study aims to provide insights into the relative benefits of yoga and walking exercise regimens on women's health, particularly in terms of body composition and metabolic health, thereby informing future exercise recommendations and health interventions.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 18-65 years； Willing and able to participate in an 8-month exercise program； Generally healthy with no contraindications to physical activity； Ability to provide informed consent

Exclusion Criteria:

Current participation in a structured exercise program； Known cardiovascular, respiratory, or metabolic disorders that contraindicate exercise； Pregnancy or planning to become pregnant during the study period； Use of medications affecting metabolism or physical activity levels； Any other condition that, in the opinion of the investigators, would make participation unsafe or not feasible

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, 8 months
  Measurement of body weight changes in kilograms from baseline to 8 months.
Change in Body Mass Index (BMI) | Baseline, 8 months
  Measurement of BMI changes calculated as weight in kilograms divided by height in meters squared from baseline to 8 months.

SECONDARY OUTCOMES:
Change in Serum Leptin Levels | Baseline, 8 months
  Measurement of serum leptin levels in ng/mL from baseline to 8 months.
Change in Fasting Blood Glucose Levels | Baseline, 8 months
  Measurement of fasting blood glucose levels in mg/dL from baseline to 8 months.
Change in Total Cholesterol (TC) Levels | Baseline, 8 months
  Measurement of total cholesterol levels in mg/dL from baseline to 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: xiaomeng liu, Principal Investigator — Zhoukou Normal University
Locations (1):
- Zhou Kou Normal University, Zhoukou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to concerns about participant privacy and the sensitivity of the health data collected.